CLINICAL TRIAL: NCT04641390
Title: Interaction Between the Vaginal and Seminal Microbiome in Patients With an Altered Vaginal Microbiome Pattern Resistant to Treatment
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Instituto Bernabeu (Other)
Responsible Party: Principal Investigator, Belen Lledo, Laboratory service manager, Instituto Bernabeu
Other Study IDs: InstitutoBernabeu2
Record Dates: First submitted 2020-11-14; First posted 2020-11-23 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Fertility Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Casos: altered vaginal microbiome resistant to drug treatment
  Interventions: Other: Analysis of the seminal microbiome of the partners of women with altered vaginal microbiome resistant to drug treatment
- Controles: Altered vaginal microbiome not resistant to drug treatment
  Interventions: Other: Analysis of the seminal microbiome of the partners of women with altered vaginal microbiome not resistant to drug treatment
- semen donors: The semen donors included in the present work will be men between 18 and 35 years old who are included in the donation program of Instituto Bernabeu after having passed a series of physical, psychological, analytical, genetic and serological evaluations and are considered suitable for donation as established by Royal Decree-Law 9/2014. Likewise, donors are subjected to a series of seminal quality evaluations and seminal freeze-thaw tests in order to guarantee their fertile potential. In this way, the donors who are part of the Instituto Bernabeu donation program also comply with current legal regulations with a strict evaluation to be considered the gold standard of potentially fertile semen. In addition, it will be necessary for them to provide a signed informed consent accepting their participation in the study.

INTERVENTIONS:
Other: Analysis of the seminal microbiome of the partners of women with altered vaginal microbiome resistant to drug treatment — The analysis of the seminal microbiome will be carried out by massive genetic sequencing
  Groups: Casos
Other: Analysis of the seminal microbiome of the partners of women with altered vaginal microbiome not resistant to drug treatment — The analysis of the seminal microbiome will be carried out by massive genetic sequencing
  Groups: Controles

SUMMARY:
It,s a retrospective case-control pilot study is to be carried out. Twenty patients will be included in the study for each branch (a total of 60). The study population will be patients whose partners have a diagnosis of an altered vaginal microbiome with (Cases, n = 20) or without (Controls, n = 20) persistence to drug treatment. Since a normal reference seminal microbiome has not been described, we will include a control group that will consist of sperm donors (n = 20) who are considered fertile potential without reproductive problems.

The main objective of the project is to identify the interaction of the vaginal and seminal microbiome patterns in couples in which the vaginal pattern is altered and is persistent to drug treatment.

ELIGIBILITY:
Inclusion Criteria:

* Woman who has an altered vaginal microbiome when the presence of bacteria of the Lactobacillus genus is less than 90% and / or the presence of bacteria that cause bacterial vaginosis (Pj: Gardnerella) or that make embryo implantation difficult in a percentage is determined greater than 5%
* Males will be between 18 and 50 years old
* Signed informed consent accepting their participation in the study.
* Male donors will be between 18 and 35 years old

Exclusion Criteria:

* Men who present with fever
* Men who are under treatment with antibiotics
* Men who have an active sexually transmitted disease
* Men who have a chronic prostatitis or a urinary infection (such as epididymitis or orchitis).

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population will be patients whose partners have a diagnosis of an altered vaginal microbiome with persistence of drug treatment or without persistence of drug treatment.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-12-15 (Estimated); Study Completion 2022-04-15 (Estimated)

PRIMARY OUTCOMES:
Participants with alteration of the vaginal microbiome resistant to drug treatment | 16 months

SECONDARY OUTCOMES:
Characteristics of the seminal microbiome of the participants whose partners with altered vaginal pattern responded well to drug treatment. | 16 months
Characteristics of the seminal microbiome pattern in patients whose partners have been diagnosed with an altered vaginal microbiome resistant to drug treatment. | 16 months
Semen donor participants eligible for donation as established by Royal Decree-Law 9/2014 to establish a seminal microbiome pattern considered optimal to compare it with participants with an altered seminal microbioma pattern. | 16 months

CONTACTS AND LOCATIONS:
Locations (1):
- University Miguel Hernández, Sant Joan d'Alacant, Alicante, Spain